CLINICAL TRIAL: NCT00916942
Title: An Open-Label Study Of The Use Of Topical Lidocaine (2.5%)/Prilocaine (2.5%) Cream As Pre-Treatment For NGX-4010 In Subjects With Postherpetic Neuralgia (PHN)
Brief Title: Study of NGX-4010 With the Use of Open Label Lidocaine (2.5%)/Prilocaine (2.5%) Cream for the Treatment of Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeurogesX (Industry)
Responsible Party: Trudy Vanhove, MD, Medical Monitor, NeurogesX
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C123
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Postherpetic Neuralgia
Keywords: Tolerability study
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Capsaicin; Lidocaine; Prilocaine

ARMS (2):
- NGX-4010 patch (Experimental)
  Interventions: Drug: capsaicin 8%
- Lidocaine (2.5%)/Prilocaine (2.5%) Cream (Experimental): Pre-treatment for NGX-4010
  Interventions: Drug: Lidocaine (2.5%)/Prilocaine (2.5%) Cream

INTERVENTIONS:
Drug: capsaicin 8% — High concentration capsaicin 8% dermal patch applied for one hour
  Arms: NGX-4010 patch
Drug: Lidocaine (2.5%)/Prilocaine (2.5%) Cream — Pre-treatment for NGX-4010
  Arms: Lidocaine (2.5%)/Prilocaine (2.5%) Cream

SUMMARY:
This study is an open-label multi-center to evaluate the tolerability of treatment with NGX-4010 use with pre-patch topical application of a topical anesthetic cream. This is an open-label study. No hypothesis testing will be performed.

Eligible subjects will have PHN and a level of pain at an intensity level deemed appropriate for open-label treatment with NGX-4010, as judged by the Investigator. Painful areas of up to a maximum of 1000 cm2 will be pre-treated with lidocaine (2.5%)/prilocaine (2.5%) cream for 60 minutes followed by a single, 60-minute application of NGX-4010. Subjects may be on chronic pain medication regimens, but currently will not be using any topical pain medications on the affected areas, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics including Lidoderm® (lidocaine patch 5%), steroids or capsaicin.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 90 years of age, inclusive.
2. Be in good health.
3. Prior diagnosis of PHN with pain persisting at least 3 months following shingles vesicle crusting.
4. Pain due to PHN that, in the opinion of the investigator, is of appropriate severity for treatment with NGX-4010. The subject should have completed at least 3 NPRS scores.
5. Intact, unbroken skin over the painful area(s) to be treated.
6. Female subjects with child-bearing potential must have a negative serum beta hCG pregnancy test, to be performed at the Screening Visit.
7. All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following study termination.
8. Be willing and able to comply with protocol requirements for the duration of study participation. (Such requirements include, but are not limited to: attending all study visits, refraining from elective surgery or extensive travel during study participation.)
9. Subjects must sign an informed consent form for this study approved by the IRB. -

Exclusion Criteria:

1. Receipt of NGX-4010 open label or blinded study patches within 12 weeks of the Study Patch Application Visit (Day 0).
2. Concomitant opioid medication, unless orally or transdermally administered and not exceeding a total daily dose of morphine 60 mg/day, or equivalent. Parenteral opioid use is excluded, regardless of dose.
3. Unavailability of an effective pain medication strategy for the subject, such as unwillingness to use opioid analgesics during study treatment, or high tolerance to opioids precluding the ability to relieve treatment-associated discomfort with oxycodone or other analgesic, as judged by the Investigator.
4. Active substance abuse or history of chronic substance abuse within the past year, or prior chronic substance abuse (including alcoholism) judged likely to recur during the study period by the investigator.
5. Recent use (within 7 days preceding the Study Patch Application Visit [Day 0]) of any topically applied pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including Lidoderm®), steroids or capsaicin products on the painful areas.
6. Current or use within the past 30 days of any investigational agent
7. Patients treated with class I (such as tocainide and mexiletine) or III anti-arrhythmic drugs.
8. Significant pain of an etiology other than PHN, for example, compression-related neuropathies (e.g., spinal stenosis), fibromyalgia or arthritis. Subjects must not have significant ongoing pain from other cause(s) that may interfere with judging PHN related pain.
9. Neuropathic pain areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes
10. Patients with congenital or idiopathic methemoglobinemia
11. Patients with glucose-6-phosphate dehydrogenase deficiencies
12. Uncontrolled (systolic blood pressure ≥ 175 mmHg or diastolic blood pressure ≥105 mmHg) or unstable hypertension
13. Clinically significant cardiovascular disease defined as cerebrovascular accident, transient ischemic attack, myocardial infarction, unstable angina, stable angina, current arrhythmia, coronary artery disease, any heart surgery including coronary artery bypass graft surgery or percutaneous coronary angioplasty/stent placement, or valvular heart disease within the past 6 months
14. Clinically significant abnormal ECG at screening.
15. Clinically significant abnormal labs at screening.
16. Significant ongoing or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function.
17. Active malignancy or past history of malignancy during the past 5 years (history of squamous cell carcinoma or basal cell carcinoma of the skin are exempted from the exclusion criteria except if they occurred in the area of treatment).
18. Any implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
19. Hypersensitivity to capsaicin (i.e., chili peppers or Over-the-Counter (OTC) capsaicin products), or any components of the capsaicin patch, Cleansing Gel, oxycodone, hydrocodone, or adhesives.
20. Patients with a known history of sensitivity to local anesthetics (including lidocaine and prilocaine) of the amide type or to any other component of the product
21. Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete daily pain diaries requiring recall of average pain level in the past 24 hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Duration of patch application | Day of treatment

SECONDARY OUTCOMES:
Mean change in NPRS scores from pre-treatment values to subsequent time points on the day of treatment | Day of treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Anchor Research Center, Naples, Florida
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Drug Studies America, Marietta, Georgia
  - A & A Pain Institute, St Louis, Missouri
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Lifetree Clinical Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Webster LR, Nunez M, Tark MD, Dunteman ED, Lu B, Tobias JK, Vanhove GF. Tolerability of NGX-4010, a capsaicin 8% dermal patch, following pretreatment with lidocaine 2.5%/prilocaine 2.5% cream in patients with post-herpetic neuralgia. BMC Anesthesiol. 2011 Dec 19;11:25. doi: 10.1186/1471-2253-11-25. PMID 22182397